CLINICAL TRIAL: NCT03413930
Title: Single-center Prospective Randomized Controlled Study of the Transanal Total Mesorectal Excision Versus Laparoscopic Total Mesorectal Excision in Rectal Cancer
Brief Title: Transanal Versus Laparoscopic Total Mesorectal Excision for Rectal Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding was raised
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Ren, Chief Physicion, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RJ-TaTME-2018
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Rectal Cancer
Keywords: TaTME; Rectal cancer; Laparoscopic Surgery
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TaTME (Experimental): Patients with mid or low rectal cancer undergo transanal total mesorectal excision.（assisted by laparoscopy to control the IMA）
  Interventions: Procedure: Transanal total mesorectal excision
- LaTME (Active Comparator): Patients with mid or low rectal cancer undergo laparoscopic total mesorectal excision.
  Interventions: Procedure: Laparoscopic total mesorectal excision

INTERVENTIONS:
Procedure: Transanal total mesorectal excision — Patients undergo transanal total mesorectal excision.（assisted by laparoscopy to control the IMA）
  Arms: TaTME
Procedure: Laparoscopic total mesorectal excision — Patients undergo Laparoscopic total mesorectal excision.
  Arms: LaTME

SUMMARY:
This study is designed to evaluate the short-term and long-term results after transanal total mesorectal excision (TaTME) for the resection of mid and low rectal cancer compared with laparoscopic total mesorectal excision（LaTME）.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) including rectal cancer is one of the most common gastrointestinal tumors, and its incidence is third in the world. At present，surgical treatments is the main means to cure CRC. Total mesorectal excision (TME) is the gold standard for rectal cancer surgery. Transanal total mesorectal excision (TaTME) was recently developed to overcome technical difficulties associated with LaTME and open TME. Most reports are retrospective studies. More studies, especially large-scale, randomized controlled trials are needed to establish the best indications for TaTME for mid and low rectal cancer.This is a single-center, open-label, non-inferiority, randomized controlled trial. A total of 120 eligible patients will be randomly assigned to TaTME group and LaTME group at a 1:1 ratio. It will provide valuable clinical evidence for the objective assessment of the oncological safety，efficacy and potential benefits of TaTME compared with LaTME for mid and low rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age < 80 years
* Body mass index (BMI) <30 kg/m2
* Tumor located in mid and low rectum ( the lower border of the tumor is located distal to the peritoneal reflection)
* Pathological rectal carcinoma
* Clinically diagnosed cT1-3N0-2 M0 lesions according to the 7th Edition of AJCC Cancer Staging Manual with or without neoadjuvant therapeutic history
* Tumor size of 5 cm or less
* ECOG score is 0-1
* ASA score is Ⅰ-Ⅲ
* Informed consent

Exclusion Criteria:

* Requiring a Mile's procedure
* Fecal incontinence
* History of inflammatory bowel disease
* Pregnant woman or lactating woman
* Severe mental disease
* Intolerance of surgery for severe comorbidities
* Previous abdominal surgery
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by rectal cancer
* Requirement of simultaneous surgery for other disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Circumferential resection margin (CRM) | 14 days after surgery
  Positive rate of circumferential resection margin (pathological assessment)

SECONDARY OUTCOMES:
Completeness of mesorectum | 14 days after surgery
  Pathological assessment of completeness of the TME specimen（complete, near
Lymph node detection | 14 days after surgery
  Lymph nodes harvested（numbers）
Distal safety margin | 14 days after surgery
  Length of distal margin （millimeter，mm）
Operative time | Intraoperative
  Operative time（minutes）
Intraoperative blood loss | Intraoperative
  Estimated blood loss（milliliters，ml）
Length of stay | 1-30 days after surgery
  Duration of hospital stay（days after surgery）
Postoperative recovery course | 1-14 days after surgery
  Time to first ambulation, flatus, liquid diet and soft diet （hours after surgery）
Early morbidity rate | 30 days
  Morbidity rate 30 days after surgery
Pain score | 1-3 days after surgery
  Postoperative pain is recorded using the visual analog scale (VAS) pain score （0-10 points）tool on postoperative day 1, 2, 3 and the day of discharge
3-year disease free survival rate | 36 months after surgery
  3-year disease free survival rate
5-year overall survival rate | 60 months after surgery
  5-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Yimei Jiang, MD, Study Chair — Ruijin Hospitla North
Locations (1):
- Ruijin Hospital North, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simillis C, Hompes R, Penna M, Rasheed S, Tekkis PP. A systematic review of transanal total mesorectal excision: is this the future of rectal cancer surgery? Colorectal Dis. 2016 Jan;18(1):19-36. doi: 10.1111/codi.13151. PMID 26466751
- [Background] Fernandez-Hevia M, Delgado S, Castells A, Tasende M, Momblan D, Diaz del Gobbo G, DeLacy B, Balust J, Lacy AM. Transanal total mesorectal excision in rectal cancer: short-term outcomes in comparison with laparoscopic surgery. Ann Surg. 2015 Feb;261(2):221-7. doi: 10.1097/SLA.0000000000000865. PMID 25185463
- [Background] Deijen CL, Velthuis S, Tsai A, Mavroveli S, de Lange-de Klerk ES, Sietses C, Tuynman JB, Lacy AM, Hanna GB, Bonjer HJ. COLOR III: a multicentre randomised clinical trial comparing transanal TME versus laparoscopic TME for mid and low rectal cancer. Surg Endosc. 2016 Aug;30(8):3210-5. doi: 10.1007/s00464-015-4615-x. Epub 2015 Nov 4. PMID 26537907